CLINICAL TRIAL: NCT04459312
Title: National Covid-Surveillance Physicians
Brief Title: National Covid-19 Surveillance Physicians
Acronym: NAT-COV-SURV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Dr. Wetzchewald (Unknown)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, Prof. Dr. Detlef Kindgen-Milles, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2020_2
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Antibody COVID-19
MeSH Terms: interventions — Antibody Formation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Antibody test (SARS-CoV2) — Antibody test

SUMMARY:
The investigators will analyze the presence of antibodies against SARS-COV2 in physicians working in emergency and intensive care medicine and in those who treat Covid 19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Qualified as physician

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All physicians working in german hospitals in emergency or intensive care medicine
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-10 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Presence of antibodies against SARS-COV2 | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Duesseldorf, Dept. of Anesthesiology, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No